CLINICAL TRIAL: NCT07265518
Title: Outpatient Induction of Labour Using a Double Balloon Transcervical Catheter in Low-risk Pregnant Women: a Two-centre Open Prospective Randomised Controlled Trial - OutCRIB
Acronym: OutCRIB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC24_0036; 2024-A02122-45 (Registry Identifier: RCB)
Record Dates: First submitted 2025-10-01; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Pregnant Women
Keywords: outpatient labor induction; low-risk pregnant women; transcervical catheter
MeSH Terms: interventions — Inosine Monophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Outpatient (Experimental): patients randomized to this arm will go home until labour or 24 hours after balloon insertion
  Interventions: Other: Outpatient
- Inpatient (Active Comparator): patients randomized to this arm will stay at hospital
  Interventions: Other: Inpatient
- observationnal study (No Intervention): patients refusing to be randomized will be able to enter this cohort without their care affecting the site's usual clinical practice

INTERVENTIONS:
Other: Outpatient — Women return at home
  Arms: Outpatient
Other: Inpatient — Women stay at hospital
  Arms: Inpatient

SUMMARY:
The aim goal of this study is to compare the duration of induction and labor between outpatient and inpatient care in low-risk pregnant women.

The secondary objectives are to compare between the two groups the maternal satisfaction from induction to delivery, the maternal and neonatal morbidity and mortality, impact on service organization and a medico-economic evaluation (cost-consequence analysis) from a collective perspective and with a time horizon of one month For women who do not agree to take part in the randomized study, an observational study will be proposed to them in order to collect the reason for their refusal and their maternal satisfaction.

Researchers will compare the return home with conventional hospitalization

Patients presenting with a singleton pregnancy and with an indication for induction of labor will be proposed to participate in the study.

If the pregnant woman refuses to participate in the randomized study, she will be invited to take part in the observational study.

For women who accept, a fetal heart rate recording (FHRR) is made prior to balloon insertion. If there is no fetal heart rhythm abnormality (FHR), the double balloon catheter is inserted by a midwife. A further ERCF is performed to ensure that the procedure is well tolerated.

In the absence of metrorrhagia, fetal heart rate abnormalities, rupture of the water sac or uterine hypertonia/hyperkinesia, the patient will then be randomized to either the in-patient or out-patient arm. The patient will either be placed in a room or go home.

In both cases, the balloon will be removed after 24 hours in hospital in the absence of spontaneous labor, and the patient will be referred to the delivery room for water breakage and/or oxytocin infusion for induction.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman with singleton pregnancy in cephalic presentation
* Term ≥ 37SA+0d
* Age ≥ 18 years
* Affiliated or beneficiary of a social security scheme
* No severe maternal/neonatal pathology (severe pre-eclampsia, intra-uterine growth retardation, etc.)
* Indication for balloon induction
* Bishop score <6
* Home-hospital distance ≤ 30 minutes' drive
* Presence of a family member at the woman's side to help her return home

Exclusion Criteria:

* Scarred uterus
* Fetal heart rhythm abnormalities
* Rupture of membranes
* Death in utero
* Placenta previa or adherent placenta (accreta or percreta)
* Maternal respiratory, cardiac, hepatic, renal, digestive or decompensated psychiatric pathology
* Anamnios
* Patient under guardianship, curatorship and/or safeguard of justice

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female gender
Enrollment: 258 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2028-01-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
compare the duration of induction and labor between outpatient and inpatient care. | 72 hours

SECONDARY OUTCOMES:
Compare maternal satisfaction from induction to delivery between the two groups outpatient and inpatient via EXIT questionnaire | 48 hours
Compare maternal morbidity and mortality between the two groups outpatient and inpatient | 48 hours
Compare neonatal morbidity and mortality between the two groups outpatient and inpatient | 48 hours
Compare the number of hospital beds freed up and the number of concurrent induction in the department | 24 hours
Compare medico-economic evaluation (cost-consequence analysis) from a collective perspective and with a time horizon of one month between the two groups outpatient and inpatient | 1 month

OTHER OUTCOMES:
Observational study: Determine patients' reasons for refusing to participate in the randomized study via an internal questionnaire | 72 hours
8. Observational study: Compare maternal satisfaction with induction between the "patients randomized to hospitalization" and "non-randomized patients (hospitalized)" groups via EXIT questionnaire | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Vincent DOCHEZ, Dr, Principal Investigator — Nantes University Hospital
Locations (2):
- France (2):
  - CHU de Nantes, Nantes, Loire Atlantique
  - CHD Vendée, La Roche-sur-Yon, vendée

IPD SHARING:
Plan to Share IPD: Undecided